CLINICAL TRIAL: NCT04808063
Title: Prevention of Incisional Hernia in Emergent Laparotomy Using a Prophylactic Mesh Augmentation Protocol Algorithm.
Brief Title: Algorithm for Prophylactic Mesh Use in Emergency Laparotomy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, Alejandro Bravo Salva, Assistant doctor, Hospital del Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CEIC2019/8240/I
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Incisional Hernia of Midline of Abdomen

STUDY DESIGN:
Intervention Model Description: Patients with emergency surgery using midline laparotomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Algorithm use for prphylactic mesh after emergency laparotomy (Experimental): Patients with emergency surgery in whom algorithm for prophylactic mesh is use to help decide abdominal wall mesh reinforcement or not.
  Interventions: Procedure: Prophylactic mesh implantation

INTERVENTIONS:
Procedure: Prophylactic mesh implantation — Use of an algorithm for prophylactic mesh implantation in high risk patients after emergency midline laparotomy.

SUMMARY:
Use of informed algorithm for patients selection of prophylactic mesh aplication after midline laparotomy in emergency surgery.

DETAILED DESCRIPTION:
Midline laparotomy complications have a high rate. When midline laparotomy is performed complications rate is even higher. One of the commons complications is incisional hernia, reaching up to 40%- 50% of cases in High risk groups.

Prophylactic mesh use has been proved to be useful preventing midline laparotomy in elective surgery. Despite this, there is not enough data to recommend its use in emergency surgery.

Aim of the study is to investigate if use of an algorithm of informed decision for use of prophylactic mesh in emergency midline laparotomy reduces incisional hernia incidence.

Prospective cohort study of all consecutive midline laparotomy performed at our emergency surgery department. Compare correct application of algorithm outcomes versus non correct application.

ELIGIBILITY:
Inclusion Criteria:

* Emergency midline laparotomy.

Exclusion Criteria:

* Surgical infection present at the moment of surgery.
* Ventrla or incisional hernia present at the moment of laparotomy .
* Open abdomen.
* Preoperative American Society of Anesthesiologist score (ASA) of V.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia | Durign first and second year of follow up
  Diagnosis by clinical or image control of incicionsal hernia during follow up.

SECONDARY OUTCOMES:
Incidence os surgical site ocurrence complications | During first postoperative month.
  Any surgical site ocurrence (SSO) complication will be registered and classified using Clavien-Dindo complication scale.
  More common complications are:
  * Seroma: a localized accumulation of serous fluid in a part of the body, occurring most commonly as a complication of a surgical procedure.
  * Wound haemathoma: wound related swelling of blood.
  * Surgical site infection: infection that occurs after surgery in the part of the body where the surgery took place. Will be classified as superficial or deep infection.
  * Wound dehiscence: lack of cutaneous healing in surgical wound.
Long term mesh related complications: chronic pain and mesh infection. | During first year of follow-up.
  Chronic pain: is any pain which persists beyond the normal healing period of 12 weeks. Visual analoge scale will be used to measure it.
  Mesh infection: Late-onset mesh infection is defined as acute inflammatory response in surgical area within months or years after operation. It is diagnosed by the presence of infection symptoms and imaging examinations.

OTHER OUTCOMES:
Global rate of complication. | Durign first month of postoperative follow up.
  Any postoperative complication will be recorded and classified using Clavien-Dindo scale.
Reintervention | During first postoperative month follow up.
  A second or subsequent intervention quotations due to postoperative comlications.
Hospital readmission | During first postoperative month follow up.
  Patient admission to a hospital within 30 days after being discharged from an earlier hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No